CLINICAL TRIAL: NCT04879030
Title: Is Combination Antibiotic Therapy Superior to Monotherapy in the Treatment of Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Combination Antibiotic Therapy Compared to Monotherapy in the Treatment of Acute COPD
Acronym: COPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPMU.01.04.21
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-02

CONDITIONS: COPD Exacerbation Acute
Keywords: COPD exacerbation; Antibiotic Therapy; beta-lactam antibiotics; fluoroquinolones
MeSH Terms: interventions — beta-Lactams; Piperacillin, Tazobactam Drug Combination; ticarcillin-clavulanic acid; Meropenem; Ertapenem; Ceftazidime; Ceftriaxone; Cefotaxime; Cefixime; Fluoroquinolones; Ciprofloxacin; Levofloxacin; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This was an open-label, randomized study using two types of treatments. Participants were divided into two groups using a randomization procedure. Within 24 hours of admission, patients were assigned randomly to two groups, one to receive a course of single-antibiotic therapy with only beta-lactam antibiotics and the other to get concomitant antibiotic treatment, defined as the use of two antibiotics, including one beta-lactam antibiotic and one fluoroquinolone. When antibiotic therapy failed, the attending physician had the right to reevaluate the clinical status and to replace the antibiotic therapy in the study with a more appropriate treatment. Patient data is stored in electronic medical records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beta-lactam monotherapy (Active Comparator): only beta-lactam antibiotics
  Interventions: Drug: Beta-Lactams
- beta-lactam and fluoroquinolone combination therapy (Experimental): one beta-lactam antibiotic and one fluoroquinolone
  Interventions: Drug: Beta-Lactams; Drug: Fluoroquinolone

INTERVENTIONS:
Drug: Beta-Lactams — The patient was randomized to use beta-lactams antibiotic
  Other Names: piperacillin-tazobactam, ticarcillin-clavulanate, imipenem-cilastin, meropenem, ertapenem, ceftazidime, ceftriaxone, cefotaxime, and cefixime
Drug: Fluoroquinolone — The patient was indicated to use a combination of beta-lactams and fluoroquinolones
  Other Names: ciprofloxacin, levofloxacin, and moxifloxacin
  Arms: beta-lactam and fluoroquinolone combination therapy

SUMMARY:
The investigators hypothesized that the empirical use of fluoroquinolones together with beta-lactam antibiotics will change their therapeutic success in patients with acute exacerbations of COPD compared to that in patients in whom a single beta-lactam treatment was used. The main goal of this study was to compare the clinical and bacterial success from the use of a combination of beta-lactam and fluoroquinolone antibiotics with that of a single beta-lactam treatment, in adult patients with COPD exacerbations.

DETAILED DESCRIPTION:
The study protocols were reviewed and approved by the Hai Phong International Hospital Institutional Review Board, Vietnam. The study was conducted in accordance with the Declaration of Helsinki and the International Conference on the Harmonization of the Technical Requirements for the Registration of Pharmaceuticals for Human Use - Good Clinical Practice guidelines. All subjects gave written informed consent before study initiation.

The participants consisted of patients aged over 45 years, diagnosed with COPD stages I-IV as stated by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 13, with acute exacerbations (onset of signs under 14 days as defined by Anthonisen et al. 14: type 1 [increased dyspnea, increased sputum volume, and sputum purulence] or type 2 [involved two or three symptoms that needed hospitalization]), the incompetence to use medication by mouth, fever (temperature over 38.5°C), antibiotic usage for longer than 1 day, treatment with systemic administration of corticosteroids (dosage equivalent to more than 30 mg of prednisolon over four days), signs of pneumonia on radiographs, history of mechanical ventilation during acute exacerbations of COPD in the past, recently detected or unresolved pulmonary malignancy, other infectious diseases requiring antibiotic treatment, and kidney failure.

Randomization and Intervention This was an open-label, randomized study using two types of treatments. Participants were divided into two groups using a randomization procedure. Within 24 hours of admission, patients were assigned randomly to two groups, one to receive a course of single-antibiotic therapy with only beta-lactam antibiotics and the other to get concomitant antibiotic treatment, defined as the use of two antibiotics, including one beta-lactam antibiotic and one fluoroquinolone. The beta-lactam antibiotics with activity against gram-negative bacilli in this study included piperacillin-tazobactam, ticarcillin-clavulanate, imipenem-cilastin, meropenem, ertapenem, ceftazidime, ceftriaxone, cefotaxime, and cefixime. The fluoroquinolone antibiotics included ciprofloxacin, levofloxacin, and moxifloxacin. The other COPD medications were continued. When antibiotic therapy failed, the attending physician had the right to reevaluate the clinical status and to replace the antibiotic therapy in the study with a more appropriate treatment. Safety was recorded daily with the support of a clinical pharmacist to report adverse events. Patient data is stored in electronic medical records.

Outcomes and Follow-Up On days 1, 10, and 20, patients were evaluated clinically, and blood was drawn, collected and the levels of C-reactive protein (CRP, Beckman Coulter Inc., Fullerton, CA) measured. Pulmonary function testing was done and expectorated sputum samples were collected. The symptoms were scored by using the visual analogue scale (VAS) for shortness of breath, tiredness, cough, and sputum color. The specific scores for each symptom ranged from 1 to 10 15. Separate and total scores were calculated.

The primary endpoint was a clinical outcome on day 20, as stated by Chow et al. 16. Successful treatment was defined as a cure (completely resolved signs and symptoms related to exacerbations) or improvement (resolved or decreased symptoms and signs without new symptoms or signs related to infection). Treatment failure was defined as the failure to address symptoms and signs, worsening of symptoms and signs, the appearance of new symptoms and signs related to the primary or a new infection, or death.

Secondary endpoints included clinical outcome on day 10 and clinical success on days 10 and 20, based on lung function (forced expiratory volume in one second [FEV1]), serum CRP, symptoms, and microbiological responses.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with COPD stages I-IV with acute exacerbations
* incompetence to use medication by mouth
* fever
* antibiotic usage for longer than 1 day
* treatment with systemic administration of corticosteroids
* signs of pneumonia on radiographs
* history of mechanical ventilation during acute exacerbations of COPD in the past

Exclusion Criteria:

* recently detected or unresolved pulmonary malignancy
* other infectious diseases requiring antibiotic treatment
* kidney failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
clinical success on day 20 | on day 20
  Proportion of patients were clinically successful on day 20 (%)
FEV1 on day 20 | on day 20
  Percent Predicted forced expiratory volume in one second on day 20 [FEV1] (%)
FVC on day 20 | on day 20
  Percent Predicted forced vital capacity (FVC) on day 20 (%)
serum CRP on day 20 | on day 20
  Concentration of serum CRP on day 20 (mg/L)
WBC on day 20 | on day 20
  white blood cell count on day 20 (10x109/L)
microbiological success on day 20 | on day 20
  The number of patients with success on microbiological outcomes on day 20
VAS on day 20 | on day 20
  the visual analogue scale (VAS) (Units on scale)
PaO2 on day 20 | on day 20
  pressure of oxygen (PaO2) on day 20 (mm Hg)
PaCO2 on day 20 | on day 20
  partial pressure of carbon dioxide (PaCO2) (mm Hg)

SECONDARY OUTCOMES:
clinical success on day 10 | on day 10
  Proportion of patients were clinically successful on day 10 (%)
FEV1 on day 10 | on day 10
  Percent Predicted forced expiratory volume in one second [FEV1] on day 10 (%)
FVC on day 10 | on day 10
  Percent Predicted forced vital capacity (FVC) on day 10 (%)
serum CRP on day 10 | on day 10
  Concentration of serum CRP on day 10 on day 10 (mg/L)
WBC on day 10 | on day 10
  white blood cell count on day 10 (10x109/L)
VAS on day 10 | on day 10
  the visual analogue scale (VAS) on day 10 (Units on scale)
PaO2 on day 10 | on day 10
  pressure of oxygen (PaO2) on day 10 (mm Hg)
PaCO2 on day 10 | on day 10
  partial pressure of carbon dioxide (PaCO2) on day 10 (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Phuong TT Nguyen, PhD MD, Principal Investigator — Haiphong University of Medicine and Pharmacy
Locations (1):
- Haiphong International Hospital, Haiphong, Vietnam

IPD SHARING:
Plan to Share IPD: No